CLINICAL TRIAL: NCT06390917
Title: Study on the Patient-Ventilator Asynchrony Analysis Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming Zhong (Other)
Responsible Party: Sponsor-Investigator, Ming Zhong, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B2024-082
Record Dates: First submitted 2024-04-18; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: To Study the Incidence of Patient-ventilator Asynchronization in Two Groups of Patients Under Two Conditions With PVA Unsynchronization Analysis Function

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With PVAs group (Experimental): With the assistance of PVA function, researchers identify the patient-ventilator asynchronies and take actions to reduce the asynchronies.
  Interventions: Device: PVA recognition function
- Without PVAs group (No Intervention): PVA function is not utilized in this arm, researchers identify the patient-ventilator asynchronies by their own and take actions to reduce the asynchronies.

INTERVENTIONS:
Device: PVA recognition function — Ventilator with the function of identify and judge PVAs
  Arms: With PVAs group

SUMMARY:
In this study, the incidence of patient-ventilator asynchronism in two groups of patients was studied when the ventilator was prompted by the PVA asynchronism analysis function

DETAILED DESCRIPTION:
Incidence of patient-computer dyssynchrony events: defined as the proportion of patient-computer dyssynchrony events in the total number of cycles during the patient trial. The observation period began 48 hours after the participants met the inclusion and exclusion criteria and signed the informed consent, and the data collection was stopped 48 hours later.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) requiring invasive mechanical ventilation
2. Patiens had spontaneous breathing;
3. Agreed to participate in the trial and signed an informed consent

Exclusion Criteria:

1. Patients with contraindications to esophageal catheter insertion and inability to monitor esophageal pressure;
2. pregnant women;
3. patients with severe central nervous system damage or neuromuscular related diseases;
4. Participating in other clinical research projects;
5. Patients deemed unsuitable by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of PVAs | 48 hours
  Percentage of the number of respiratory cycles in which human-machine asynchronous events occurred in the total number of respiratory cycles in each patient during the trial

SECONDARY OUTCOMES:
The proportion of PVAs that were identified by the investigator among the total PVAs during the trial | 48 hours
Incidence of PVA within half an hour before and after the intervention | Half an hour before and after the intervention
Accuracy of PVA recognition function | 48 hours
  Compare manual audit and machine judgment

IPD SHARING:
Plan to Share IPD: Undecided